CLINICAL TRIAL: NCT00762320
Title: Comparison of Liquid Kaletra and Low Dose Kaletra Tablets in HIV-Positive Children
Brief Title: Comparison of Liquid Kaletra and Low Dose Kaletra Tablets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phoenix Children's Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Janice Piatt, Medical Director, Bill Holt Clinic, Phoenix Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-017
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Results first posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-02

CONDITIONS: HIV Infections
Keywords: HIV; Kaletra; treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — lopinavir-ritonavir drug combination; Lopinavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low dose Kaletra tablets (Experimental): Patients will serve as their own controls as they are switched from the baseline treatment with liquid Kaletra to the study intervention treatment with Low Dose Tablet Kaletra (100mg/25mg)
  Interventions: Drug: Low dose Kaletra tablets

INTERVENTIONS:
Drug: Low dose Kaletra tablets — Lopinavir/Ritonavir tablets 100mg/25mg
  Other Names: lopinavir/ritonavir 100mg/25mg

SUMMARY:
Kaletra (a combination drug with lopinavir and ritonavir) is one of a few effective medications that are approved and available for young children who are HIV+. The liquid form is reported to have a very nasty taste and presents difficulties for the children who must take the medication twice a day and for their parents who must enforce the medication regimen. The children are often well into their teens before they weigh enough to be able to take the adult dose tablet (200mg/50mg). A new smaller dose tablet (100mg/25mg) is now available. However, it is not known if the liquid and tablet act the same in children. The purpose of this study is to switch children from the baseline treatment with the liquid to the study intervention treatment with 100mg/25mg tablet form of Kaletra. The study will compare children pre-switch and post-switch in terms of how well their HIV is controlled . Comparisons of parent and child satisfaction will also be made. Eight to 10 HIV+ children currently well managed with a medications including liquid Kaletra will be invited to switch from the liquid to the low dose Kaletra tablet. The parent and/or child will complete a satisfaction survey for the liquid Kaletra and lab values will be taken from the chart. At the time of the switch and 1, 3 and 6 months post switch blood tests will be drawn and the parent and/or child will complete the satisfaction survey. In addition, at the switch and 1 month post switch, a day will be spent in clinic with 5 blood draws to see how much of the drug is in the blood stream at different times after the medicine is taken.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ children aged 3-18.
* Baseline treatment includes liquid Kaletra
* currently on a stable (on same regimen > 3 months, Viral Load< 5,000), Highly Active Antiretroviral Therapy (HAART) regimen
* able to take pills or willing to undergo pill training prior to enrollment
* weight must be greater than or equal to 15kg

Exclusion Criteria:

* Unable to swallow pills
* Concomitant treatment with Rifampin or St. John's Wort which have been shown to decrease plasma concentrations of lopinavir.
* Concurrent use of drugs primarily metabolized by CYP3A, which metabolizes ritonavir: Astemizole, Cisapride, Dihydroergotamine, Ergonovine, Ergotamine, Flecainide, Lovastatin, Methylergonovine, Midazolam, Pimozide, Propafenone, Simvastatin, terfenadine, Triazolam
* Baseline treatment does NOT include Kaletra

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Piatt, MD, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients weighing 15kg and able to swallow pills, currently taking liquid lpv/rtv were recruited from an outpatient pediatric HIV clinic from 4/1/2009 through 1/12/11
Groups:
- Low Dose Kaletra: Patients will serve as their own controls as they are switched from liquid Kaletra to Low Dose Tablet Kaletra
  Low dose Kaletra tablets : Lopinavir/Ritonavir tablets 100mg/25mg
Period: Overall Study
Arm/Group | Low Dose Kaletra
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Low Dose Kaletra
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.18 (1.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Absolute CD4 and CD4 %
Description: Number of participants who had no clinically significant deterioration in absolute CD4 and % CD4 count for the duration of the study. Absolute CD4 and Percent CD4 counts were determined by single or dual platform analysis performed on blood samples by Phoenix Children's Hospital Laboratory, Sonora Quest Laboratory or Labcorp Laboratory. Clinically significant change was determine to be a deterioration in both Absolute CD4 to less than 500 and %CD4 to less than 25%.
Time Frame: Baseline, 4 weeks, 12 weeks, 26 weeks
Population: All participants were analyzed.
Measure: Number; unit: participants
Groups:
- Low Dose Kaletra: Patients receiving Low Dose Kaletra Tablets
Arm/Group | Low Dose Kaletra
Number analyzed (Participants) | 8
participants | 8

2. Primary Outcome: Lopinavir (Lpv) and Ritonavir (Rtv) Maximumu Plasma Concentration (CMax) Liquid
Description: Cmax values at baseline (participants are taking liquid Kaletra as part of baseline treatment). Time points for data collection: 0, 2hrs post dose, 4 hrs post dose, 8 hrs post dose.
Time Frame: Baseline
Population: All participants were analyzed
Measure: Median (Standard Deviation); unit: ng/ml
Arm/Group | Low Dose Kaletra
Number analyzed (Participants) | 8
ng/ml
  Cmax Lpv | 9742 (2533.9)
  Cmax Rtv | 637.0 (357.5)

3. Primary Outcome: Lopinavir and Ritonavir Area Under the Curve (AUC) Liquid Kaletra
Description: Area under the curve values for lopinavir at baseline when participants are taking liquid Kaletra as part of their baseline treatment. Time points for data collection: 0, 2 hrs post, 4 hrs post, 6 hrs post, 8 hrs post.
Time Frame: Baseline
Population: All participants were analyzed
Measure: Median (Standard Deviation); unit: hr*ng/ml
Arm/Group | Low Dose Kaletra
Number analyzed (Participants) | 8
hr*ng/ml
  Lpv AUC at baseline | 90651 (30346.4)
  Rtv AUC at baseline | 3701.2 (2088.0)

4. Primary Outcome: Lopinavir AUC Ratio of Baseline:Week 4
Description: Ratio of AUC at baseline (liquid)to week 4 (reduced dose tablet). AUC data were collected at 0, 2, 4, 6, and 8 hours post dose.
Time Frame: Baseline, week 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Low Dose Kaletra
Number analyzed (Participants) | 8
ratio | 1.01 (.36)

5. Secondary Outcome: Patient Satisfaction
Description: Patient Satisfaction Survey. Eight item Likert scale of patient satisfaction with their HIV treatment regimen for patients 7 years of age and older. Items scores are summed to compute a total score. Total scores are reported with a minimum of 0 and a maximum of 32, with higher scores indicating higher satisfaction.
Time Frame: Baseline, 1 month
Population: Patients had to be able to read and write to complete the patient satisfaction questionnaire, so an arbitrary age of 7 was selected and patients under the age of 7 did not complete the patient satisfaction questionnaire. All 5 of the patients over the age of 5 completed the questionnaire and were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Low Dose Kaletra Baseline Visit: Patient satisfaction score at baseline visit
- Low Dose Kaletra Week 4 Visit: Patient Satisfaction Score at Week 4 visit
Arm/Group | Low Dose Kaletra Baseline Visit | Low Dose Kaletra Week 4 Visit
Number analyzed (Participants) | 5 | 5
units on a scale | 20.2 (7.76) | 21.8 (6.02)
Statistical Analysis 1: Comparison: Low Dose Kaletra Baseline Visit vs Low Dose Kaletra Week 4 Visit; Test type: Superiority or Other; p = .004, t-test, 2 sided; df=4

6. Secondary Outcome: Symptoms Across All Patients
Description: Cumulative tally of symptoms for each patients across all visits. Targetted symptoms were asked for at each visit and patients and parents were encouraged to report additional symptoms that were experienced. Each patient got a score for the total number of symptoms at each visit. Scores were totalled, but it the same symptoms occurred continuously it was counted as 1 symptom.
Time Frame: Baseline, 1 month, 3 months, 6 months
Population: All participants analyzed
Measure: Mean (Standard Deviation); unit: numer of symptoms
Groups:
- Low Dose Kaletra: Patients receiving Low Dose Kaletra
Arm/Group | Low Dose Kaletra
Number analyzed (Participants) | 8
numer of symptoms
  Symptoms for all subjects at Baseline | 20.20 (7.76)
  Symptoms for all subjects at 4 Weeks | 21.80 (6.02)
  Symptoms for all subjects at 12 Weeks | 26.40 (2.30)
  Symptoms for all subjects at 24 weeks | 26.60 (3.21)

7. Primary Outcome: Viral Load (VL)
Description: Number of participants who maintained their Viral load undetectable (< 20 copies/ml) for the duration of the study
Time Frame: Baseline, Week 4, Week 12 and Week 24
Population: All subjects in study were analyzed
Measure: Number; unit: participants
Arm/Group | Low Dose Kaletra
Number analyzed (Participants) | 8
participants | 8

8. Primary Outcome: Lopinavir (Lpv) and Ritonavir (Rtv) Cmax at 4 Weeks
Description: Lpv and rtv Cmax at 4 weeks when participants are receiving study intervention, low dose Kaletra. Time points for data collection: 0, 2hrs, 4hrs, 6hrs, 8hrs
Time Frame: 4 weeks
Population: All participants were analyzed
Measure: Median (Standard Deviation); unit: ng/ml
Arm/Group | Low Dose Kaletra
Number analyzed (Participants) | 8
ng/ml
  Lpv Cmax at 4 weeks | 11143 (2839.5)
  Rtv Cmax at 4 weeks | 912.1 (588.9)

9. Primary Outcome: Lopinavir and Ritonavir AUC on Low Dose Tablet
Description: Lopinavir and Ritonavir AUC at 4 weeks when participants are receiving the study intervention, low dose tablet formulation of Kaletra. Data collection points for AUC were 0, 2, 4, 6, and 8 hours post dose.
Time Frame: 4 weeks
Population: All participants were analyzed
Measure: Median (Standard Deviation); unit: hr*ng/ml
Arm/Group | Low Dose Kaletra
Number analyzed (Participants) | 8
hr*ng/ml
  Lpv AUC at 4 weeks | 85670 (25184.5)
  Rtv AUC at 4 weeks | 4876.1 (2541.0)

10. Secondary Outcome: Parent Satisfaction
Description: Parent Satisfaction Survey. Eight item Likert scale of parent/guardian satisfaction with the child's HIV treatment regimen. Item scores are summed to compute a total score. Total scores are reported with a minimum of 0 and a maximum of 32, with higher scores indicating higher satisfaction.
Time Frame: Baseline, 4 week, 12 weeks and 24 weeks
Measure: Mean (Standard Deviation); unit: Score on a survey
Groups:
- Low Dose Kaletra Baseline: Patients receiving Low Dose Kaletra at baseline
- Low Dose Kaletra Week 4: Patients Receiving Low Dose Kaletra at Week 4
Arm/Group | Low Dose Kaletra Baseline | Low Dose Kaletra Week 4
Number analyzed (Participants) | 8 | 8
Score on a survey | 26.75 (3.92) | 28.38 (3.02)
Statistical Analysis 1: Comparison: Low Dose Kaletra Baseline vs Low Dose Kaletra Week 4; Test type: Superiority or Other; p < .001, t-test, 2 sided; df=7

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 24 weeks after switch from liquid to low dose tablet formulation of Kaletra
Arm/Group | Low Dose Kaletra
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Kaletra (N=8)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Pain due to previously scheduled orthopedic surgery
Throat Pain (General disorders) | 1 (4)
fever (General disorders) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (8)
anorexia (Gastrointestinal disorders) | 1 (1)
ear pain (Ear and labyrinth disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 4 (4)
nausea (Gastrointestinal disorders) | 2 (3)
headache (General disorders) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (8)
difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 3 (6)
leg pain (Musculoskeletal and connective tissue disorders) | 2 (7) — leg cramps or leg pain
leg fatigue (Musculoskeletal and connective tissue disorders) | 1 (2)
Increased MCV (Investigations) | 7 (23)
Increased Cholesterol (Investigations) | 7 (24)
Increased Triglycerides (Investigations) | 2 (3)
increased amylase (Investigations) | 5 (8)
Increased Monocytes (Investigations) | 1 (1)
Increased WBC (Investigations) | 2 (2)
decreased RBC (Investigations) | 4 (8)
decreased plt (Investigations) | 2 (2)
Increased eosinophils (Investigations) | 4 (4)
decreased neutrophil percent (Investigations) | 3 (7)
decreased ANC (Investigations) | 2 (4)
Increased lymphocyte percent (Investigations) | 3 (8)
increased HCT (Investigations) | 1 (1)
decreased CO2 (Investigations) | 2 (2)
increased CO2 (Investigations) | 1 (1)
Increased Alk Phos (Investigations) | 1 (2)
Decreased Na+ (Investigations) | 1 (1)
Increased K+ (Investigations) | 1 (1)
decreased K+ (Investigations) | 1 (1)
Increased Creatinine (Investigations) | 1 (2)

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No